CLINICAL TRIAL: NCT04839939
Title: Short Term Efficacy of Combination Taping Technique as an Alternative to Ankle Foot Orthosis on Improving Gait Parameters in Spastic Cerebral Palsy: A Controlled Randomized Study
Brief Title: Efficacy of Combination Taping Technique vs Ankle Foot Orthosis on Improving Gait Parameters in Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Batterjee Medical College (Other)
Collaborators: Taif University (Other)
Responsible Party: Principal Investigator, Mohamed A. Abdel Ghafar, Associate Professor, Batterjee Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Batterjee
Record Dates: First submitted 2021-03-31; First posted 2021-04-09 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Gait; Spastic Diplegia
Keywords: Combination Taping; Ankle foot orthosis; Spatio-temporal paremeters
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Active Comparator): Children in this group received conventional physical therapy program in form of Stretching for tight muscles, weak muscles Strengthening, Postural reactions training, Proprioceptive training, and Walking training were all part of the treatment plan, which was based on the neurodevelopmental approach.
  Interventions: Other: Conventional physical therapy
- AFO Group (Experimental): Children in this group received the same conventional treatment plus they were provided with solid community-prescribed AFO with a wearing schedule of 6-12 hours per day. Parents were given a detailed demonstration about how to use the AFO probably and watching for areas of skin overpressure. AFO needs to be worn with a smooth, long sock underneath with the child's heel is right down in the AFO with the ankle strap and/or shoe fastened firmly.
  Interventions: Other: Ankle Foot Orthosis
- Combination Taping Group (Experimental): Children in this group received the same conventional treatment plus the combination taping technique, which was performed by one qualified physical therapist with over five years of experience. The technique started with the application of two 5-cm wide Kinesio tape "I" straps. The first strap was applied from the lateral condyle of the tibia to the base of the first metatarsal bone with the ankle joint in plantar flexion. The tape was not stretched for 5 cm from the initial site and was then stretched up to 30% for the remaining parts15. The second "I" strap While the therapist holds the ankle in dorsiflexion, he applied the distal end of the tape 10 cm below the ankle joint. With almost 70% tension, the proximal end is applied 10 cm above the ankle joint. While one hand was holding each end of the tape, the child was asked to move the joint into plantar flexion. Finally, both hands moved towards the middle of the joint to apply the remaining tape.
  Interventions: Other: Combination Taping

INTERVENTIONS:
Other: Conventional physical therapy — Stretching for tight muscles, weak muscles Strengthening, Postural reactions training, Proprioceptive training, and Walking training
  Arms: Control Group
Other: Ankle Foot Orthosis — Solid prescribed AFO with a wearing schedule of 6-12 hours per day
  Arms: AFO Group
Other: Combination Taping — Combination between elastic and inelastic taping
  Arms: Combination Taping Group

SUMMARY:
Gait in children with spastic CP is often characterized by abnormal gait kinematics as knee flexion and equines foot which associated with such gait deviations, an elevated walking energy cost is often observed which may contribute to activity limitations.

The ability to maintain proper joint alignment of the lower extremity, and control the position of the foot in standing and walking is a critical treatment objective for gait in children with cerebral palsy. Lower extremity orthoses, such as ankle-foot orthoses (AFOs) are widely recommended in children with spastic cerebral palsy to prevent the development or progression of this deformity and to improve the dynamic efficiency of the child's gait. The use of Kinesio taping in pediatric rehabilitation becomes increasingly popular in recent years. Recent systematic reviews reported moderate evidence that Kinesiology taping is a useful adjunct to physiotherapy intervention in higher functioning children with CP. Combination tapings is a technique first introduced by Kenzo Kase, in which Kinesio taping is coupled with the rigid athletic tape to maximize the treatment benefits. This approach remains briefly addressed in the literature with no prior studies has examined the effects of combination tapings in the CP pediatric population. Hypothesis: there is no difference between the effect of combining tapings and ankle-foot orthosis on spatiotemporal gait parameters in spastic cerebral palsied

DETAILED DESCRIPTION:
This study was designed as a randomized controlled trial. The participants and their parents were given clear, detailed explanation of the proposed procedures before starting the experiment, and signed a written informed consent statement. Batterjee Medical College Research and Ethical committee reviewed and approved the study, which were conducted in compliance with the 1975 Helsinki Declaration. Thirty-six children (22 males and 14 females) with spastic diplegic cerebral palsy were enrolled in this study. The children were randomly assigned into two study groups (A & B), and a control group (C). Randomization was done by asking each child to pick up an index card out of a box that contains 36 cards (12 cards for each group) to determine which group participants would be in. Measurements were taken in two occasions, baseline, and four weeks after application of the intervention. Spatiotemporal Gait parameters were measured as per the published guidelines using the GAITRite system. Parameters included were cadence, step length; stride length, single support time, double support time, and velocity were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age range from 8 to 15 years old
* Able to stand and walk independently
* Spasticity ranged from 1 to 1+ grade according to Modified Ashworth Scale
* level I or II according to Gross Motor Function Classification System (GMFCS)
* Able to understand and follow instructions

Exclusion Criteria:

* Children with previous corrective orthopedic surgery or botulinum toxin injection in the lower extremities within the previous 6 months
* Skin disease
* Epilepsy
* Mental retardation
* Visual or auditory problems

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Step Length (cm) | 4 Weeks
  Change of the step length was measured using GAITRite System
Stride Length (cm) | 4 Weeks
  Change of the stride length was measured using GAITRite System
Velocity (cm/s) | 4 weeks
  Change of the velocity was measured using GAITRite System
Cadence (step/min) | 4 weeks
  Change of the cadence was measured using GAITRite System
Single leg support (% of gait cycle) | 4 weeks
  Change of the single leg support was measured using GAITRite System
Double leg support (% of gait cycle) | 4 weeks
  Change of the double leg support was measured using GAITRite System

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed M. Abdel Ghafar, Ph.D, Principal Investigator — Batterjee Medical College
Locations (1):
- Fizik Center For Physiotherapy, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No